CLINICAL TRIAL: NCT03839147
Title: The Effect of Education and Counseling on Reducing Pain and Anxiety in Women Undergoing Hysterosalpingography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 50687469
Record Dates: First submitted 2019-02-07; First posted 2019-02-15 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2019-02

CONDITIONS: Women's Health
Keywords: hysterosalpingography; anxiety; pain; education; counseling
MeSH Terms: conditions — Anxiety Disorders; Pain | interventions — Educational Status; Counseling

STUDY DESIGN:
Intervention Model Description: This randomized controlled study was conducted at Gulhane Training and Research Hospital, Obstetrics and Gynecology clinic between May 2016 and January 2017. The CONSORT (Consolidated Standards of Reporting Trials) guidelines for reporting randomised controlled trials (RCTs) has been used to describe the methods.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education and Counseling (Experimental): After obtaining written informed consent, the data collection form, Spielberger State Anxiety Scale and visual analogue scale scoring scale were applied to both groups by face to face interview during the day giving appointment for hysterosalpingography. Immediately after the questionnaires were applied, the nurse gave individual education and counseling were giving by the nurse researcher to intervention group for 30 minutes. This education consisted of the definition and the purpose of hysterosalpingography, when and how it was applied, in what cases it was applied, whether it was a painful procedure, possible side effects and additional benefits of infertility treatment
  Interventions: Behavioral: Education and counseling
- Control group (No Intervention): Participants in the control group received standard care (verbal information about procedure and a short written information about the procedure) and no intervention (education and counseling) was performed. Both groups were re-evaluated using the same scales after the hysterosalpingography. Within 5 minutes of completing the hysterosalpingography procedure, participants were asked to evaluate their pain in order to characterize pain intensity using the visual analogue scale .

INTERVENTIONS:
Behavioral: Education and counseling — After obtaining informed consent, the data collection form, Spielberger State Anxiety Scale and VAS scoring scale were applied to both groups by face to face interview during the day giving appointment for HSG. Immediately after the questionnaires were answered, individual education and counseling were giving by the nurse researcher to intervention group for 30 minutes. In addition, the education and counseling given to the participants by the researcher was repeated briefly on the morning of the HSG procedure and any questions of the patients were answered.
  Arms: Education and Counseling

SUMMARY:
This study investigates the effect of education and counseling on anxiety and pain in women undergoing hysterosalpingography as part of the infertility process.

DETAILED DESCRIPTION:
Fertility and having a child is a significant experience for most individuals; however, many struggle to achieve pregnancy. Infertility is defined as the inability of a couple to conceive after 12 months of regular unprotected sexual intercourse or to carry a pregnancy to term. It is estimated that 10-15 % of the couples globally experience infertility. In Turkey, it is estimated that 10-20% of the couples are diagnosed with infertility. In the evaluation of infertile couples, hysterosalpingography (HSG) is a simple, safe, and minimally invasive radiologic procedure to visualize uterine cavity and tubes after contrast enhancement. HSG plays an important diagnostic role in finding the cause of infertility and in deciding the line of management. The aim of this study was to investigate the effect of education and counseling on anxiety and pain before the treatment of women who will have HSG procedure with the diagnosis of infertility.

This randomized controlled study was conducted at Gulhane Training and Research Hospital, Obstetrics and Gynecology clinic between May 2016 and January 2017. Volunteer women undergoing HSG as part of infertility evaluation have been included. Participants were randomly assigned to the intervention or the control group using a computer-generated list. A data collection form including socio-demographic and obstetric characteristics such as age, educational status, duration of infertility, previous pregnancies, births, abortion/curettage numbers, Spielberger State Anxiety Scale and Visual Analog Scale scores was used for each patient. After obtaining written informed consent, the data collection form, Spielberger State Anxiety Scale and VAS scoring scale were applied to both groups by face to face interview during the day giving appointment for HSG. Immediately after the questionnaires were applied, the nurse gave individual education and counseling were giving by the nurse researcher to intervention group for 30 minutes. Participants in the control group received standard care (verbal information about procedure and a short written information about the procedure) and no intervention (education and counseling) was performed.The IBM SPSS (Statistical package for the Social Sciences) 22.0 package program was used to evaluate the data obtained in the study.

ELIGIBILITY:
Inclusion Criteria:

* being diagnosed with infertility
* negative the result of the B-HCG testing
* being able to understand, read and write in Turkish

Exclusion Criteria:

* not wanting to be included in the study
* not accepting education/counseling
* not knowing Turkish
* having additional diseases related to pelvic pain

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 105 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Spielberger State Anxiety Scale | 30 minutes
  After completing the HSG procedure, participants filled out the Spielberger State Anxiety Scale.
  The Spielberger state anxiety scale was developed in 1964 by Spielberger. There are 20 statements in the scale that individuals can use to express their feelings. The State Scale measures the level of anxiety related to the situation and has been scored by four options for each expression. These are: "None" (1), "Slightly" (2), "Many" (3), "Completely" (4). The statements in this section are divided directly and reversed. Reversed statements are 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20.
  The total score of the expressions which are reversed from the total score of the direct expressions and adding the number 50 which is the constant value of the state anxiety scale. Spielberger and his colleagues stated that 0-19 points obtained from the scale meant "no anxiety", 20-39 points meant "light", 40-59 points meant "medium", 60-79 points meant "heavy anxiety".
Visual Analog Scale for pain intensity | 10 minutes
  After completing the HSG procedure, participants were asked to evaluate their pain in order to characterize pain intensity using the Visual Analog Scale (VAS). Patients indicated the maximum pain intensity experienced during the HSG by making a vertical line on the VAS.
  A standard ten-point visual analogue scale (VAS) of 0 to 10 was designed and used to assess the patients' perceptions of discomfort during the procedure. A high score on the scale indicated a high level of discomfort and a score of 0 denoted no discomfort at all. Patients indicate the degree of pain they feel between 0-10.

CONTACTS AND LOCATIONS:
Overall Officials: Gulten Guvenc, Principal Investigator — University of Health Sciences, Gulhane Faculty of Nursing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aba YA, Avci D, Guzel Y, Ozcelik SK, Gurtekin B. Effect of music therapy on the anxiety levels and pregnancy rate of women undergoing in vitro fertilization-embryo transfer: A randomized controlled trial. Appl Nurs Res. 2017 Aug;36:19-24. doi: 10.1016/j.apnr.2017.05.005. Epub 2017 May 22. PMID 28720234
- [Background] Onwuchekwa CR, Oriji VK. Hysterosalpingographic (HSG) Pattern of Infertility in Women of Reproductive Age. J Hum Reprod Sci. 2017 Jul-Sep;10(3):178-184. doi: 10.4103/jhrs.JHRS_121_16. PMID 29142446
- [Result] Stevenson EL, Hershberger PE, Bergh PA. Evidence-Based Care for Couples With Infertility. J Obstet Gynecol Neonatal Nurs. 2016 Jan-Feb;45(1):100-10; quiz e1-2. doi: 10.1016/j.jogn.2015.10.006. Epub 2015 Dec 1. PMID 26815804